CLINICAL TRIAL: NCT07060365
Title: A Master Protocol Phase I/II Study to Investigate Biomarker-Guided Novel Anticancer Agent(s) as Monotherapy or Combination Therapy for the Treatment of Participants With Advanced/Recurrent Ovarian Cancer (Ovarian Platform)
Brief Title: A Master Protocol Study to Investigate Biomarker-guided Novel Anticancer Agent(s) as Monotherapy or Combination Therapy in Participants With Advanced/Recurrent Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9724C00001
Record Dates: First submitted 2025-06-24; First posted 2025-07-11 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Advanced/Recurrent Ovarian Cancer
Keywords: Novel Anticancer Agent; Biomarker-Guided; Novel PARPi; BRCA1/2m; Neoadjuvant treatment
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Saruparib (Experimental): Participants will receive saruparib via oral administration.
  Interventions: Drug: Saruparib

INTERVENTIONS:
Drug: Saruparib — Participants will receive saruparib via oral administration.

SUMMARY:
The main purpose of this study is to investigate the safety, tolerability, preliminary efficacy, pharmacokinetics (PK) and pharmacodynamics (PD) of biomarker-guided novel anticancer agent(s) as monotherapy or combination therapy for the treatment of participants with advanced/recurrent ovarian cancer.

Substudy 1 will investigate the safety, tolerability, preliminary efficacy, PK and PD of saruparib monotherapy in participants with BReast CAncer gene (BRCA) mutated epithelial ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
This Phase I/II, open-label, multicentre study will employ a platform design utilising a Master Protocol with multiple parallel, open-label substudies.

Substudy 1 is a single-arm, open label, Phase II multicentre study investigating the safety, tolerability, preliminary efficacy, PK, and PD of saruparib monotherapy, as neoadjuvant treatment in participants with newly diagnosed, tBRCA1/2m International Federation of Gynecology and Obstetrics (FIGO) 2014 Stage III/IV epithelial ovarian, fallopian tube, or primary peritoneal cancer, and who are eligible for neoadjuvant treatment with planned interval debulking surgery (IDS).

ELIGIBILITY:
Key Inclusion Criteria:

Master Protocol:

1. Participants who have histologically or cytologically documented advanced or recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer, considered to be suitable for treatment with study intervention, as applicable to each substudy.
2. Participants must provide sufficient archival or fresh tumour sample for biomarker testing.
3. Life expectancy at the time of screening ≥ 12 weeks in the opinion of the Investigator.
4. Measurable disease as per RECIST 1.1 criteria: at least one lesion that can be accurately measured at baseline as ≥ 10 mm in the longest diameter.
5. ECOG PS of 0 to 1, with no deterioration over the previous 2 weeks prior to baseline at screening, and prior to study intervention administration.
6. Adequate organ and marrow function.

Substudy 1:

1. Participants must have histologically or cytologically confirmed newly diagnosed FIGO 2014 Stage III/IV epithelial ovarian*, fallopian tube, or primary peritoneal cancer who are eligible for neoadjuvant treatment with planned IDS.
2. Participants who are treatment-naïve.
3. Participants with evidence of predicted loss of function tBRCA1/2m (by local testing) as assessed by a commercially available diagnostic test.

Key Exclusion Criteria:

Master Protocol:

1. Any history of persisting (> 2 weeks) severe pancytopenia due to any cause (absolute neutrophil count < 0.5 × 10/Liters (L) or platelets < 50 × 10/L).
2. Spinal cord compression or brain metastases unless asymptomatic, treated, and stable and not requiring continuous corticosteroids prednisone/day or dexamethasone or equivalent for at least 4 weeks prior to start of study intervention. Participants with leptomeningeal carcinomatosis are excluded.
3. Active primary immunodeficiency/active infectious disease(s).
4. Participants with any known predisposition to bleeding (eg, active peptic ulceration, recent [within 6 months] haemorrhagic stroke, proliferative diabetic retinopathy).
5. Cardiac criteria, including history of arrhythmia and cardiovascular disease.
6. Prior malignancy that required treatment within 2 years prior to screening.
7. Previous allogeneic bone marrow or solid organ transplant.
8. As judged by the Investigator, any evidence of severe or uncontrolled systemic diseases or active uncontrolled infections.
9. Known allergy or hypersensitivity to investigational product(s) or any of the excipients of the investigational product(s) (as applicable to a substudy).
10. Concomitant use of drugs that are known to prolong or shorten QT and have a known risk of (Torsades de Pointes) TdP.
11. During the 4 weeks prior to the first dose, receiving continuous corticosteroids prednisone/day or equivalent for any reason.
12. Major surgical procedure (excluding placement of vascular access) or significant traumatic injury.
13. Any concurrent anticancer therapy.

Substudy 1:

1. Participants with history of myelodysplastic syndrome (MDS) or acute myeloid leukaemia (AML) or with features suggestive of MDS/AML (as determined by prior diagnostic investigation). Specific screening for MDS/AML is not required.
2. Refractory nausea and vomiting, clinical signs or symptoms of Gastrointestinal (GI) obstruction and/or requirement for parenteral hydration or nutrition, history of prior intestinal obstruction, chronic GI diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of saruparib.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2029-03-27 (Estimated); Study Completion 2029-03-27 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse event (TEAEs), serious adverse events (SAEs), and adverse events (AEs) leading to discontinuation | From Day 1 to Survival Follow up (approximately 6 months)
  To assess the safety and tolerability of novel biomarker guided treatment in participants with advanced/recurrent ovarian cancer.

SECONDARY OUTCOMES:
Substudy 1: Estimate of objective response rate (ORR) defined as proportion of participants who have a complete or partial response | From Day 1 to IDS surgery (within 6 weeks after conclusion of study intervention treatment [Day 1 until 12 weeks])
  To estimate the efficacy of neoadjuvant treatment (and prior to IDS) with saruparib single-agent by assessment of ORR in participants with newly diagnosed tBRCA1/2m advanced epithelial ovarian cancer and with measurable disease at baseline.
Substudy 1: Estimate of confirmed cancer antigen 125 (CA125) response rate defined as at least 50% reduction in serum CA-125 levels from pre-treatment levels | Screening (Day -28), Day 1 (Cycle 1) and Day 15 (Cycle 2) (28-day cycles), End of Treatment (7 days after final dose), Pre-surgery Follow up
  To estimate the efficacy of neoadjuvant treatment (and prior to IDS) with saruparib single-agent in participants with newly diagnosed tBRCA1/2m advanced epithelial ovarian cancer and evaluable for CA125 response per the GCIG criteria.
Substudy 1: Proportion of participants with pathological complete response (pCR) defined as no macroscopic residual and no microscopic (viable) disease on histologic evaluation of all surgical specimens | IDS Follow up period (IDS surgery within 6 weeks after conclusion of study intervention treatment [Day 1 until 12 weeks])
  To estimate the efficacy of neoadjuvant treatment with saruparib single-agent by assessment of pCR in participants with newly diagnosed tBRCA1/2m advanced epithelial ovarian cancer and with measurable disease at baseline.
Substudy 1: Proportion of participants with complete surgical resection of tumour at IDS defined as no macroscopic tumour remains after surgery | IDS Follow up period (IDS surgery within 6 weeks after conclusion of study intervention treatment [Day 1 until 12 weeks])
  To estimate the efficacy of neoadjuvant treatment with saruparib single-agent by assessment of CRR in participants with newly diagnosed tBRCA1/2m advanced epithelial ovarian cancer and with measurable disease at baseline.
Substudy 1: Area under the plasma drug concentration-time curve (AUC) | Day 1 (Cycle 1 and Cycle 3) (28-day cycles)
  To characterise the PK of saruparib and its metabolite(s) if applicable, as monotherapy in plasma following a single dose and at steady state after multiple dosing, when given orally as neoadjuvant monotherapy prior to IDS participants with newly diagnosed tBRCA1/2m advanced epithelial ovarian cancer.
Substudy 1: Maximum plasma concentration of the drug (Cmax) | Day 1 (Cycle 1 and Cycle 3) (28-day cycles)
  To characterise the PK of saruparib and its metabolite(s) if applicable, as monotherapy in plasma following a single dose and at steady state after multiple dosing, when given orally as neoadjuvant monotherapy prior to IDS participants with newly diagnosed tBRCA1/2m advanced epithelial ovarian cancer.
Substudy 1: Time to maximum plasma concentration (tmax) | Day 1 (Cycle 1 and Cycle 3) (28-day cycles)
  To characterise the PK of saruparib and its metabolite(s) if applicable, as monotherapy in plasma following a single dose and at steady state after multiple dosing, when given orally as neoadjuvant monotherapy prior to IDS participants with newly diagnosed tBRCA1/2m advanced epithelial ovarian cancer.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (5):
  - Research Site, Fullerton, California
  - Research Site, Albuquerque, New Mexico
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Seattle, Washington
- Italy (4):
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Ravenna
  - Research Site, Rome
- South Korea (2):
  - Research Site, Goyang
  - Research Site, Seoul
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosuree.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/